CLINICAL TRIAL: NCT06911723
Title: Activities to Change Your Mood: A Test of the Acceptability and Initial Efficacy in Clinical Samples and Healthy Controls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lauren Luther, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300014130; Internal Award (Other Grant/Funding Number: University of Alabama at Birmingham)
Record Dates: First submitted 2025-03-18; First posted 2025-04-04 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia Disorders
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Coping Activities (Experimental)
  Interventions: Behavioral: Brief Activities
- Belief Modifying Activities (Experimental)
  Interventions: Behavioral: Brief Activities

INTERVENTIONS:
Behavioral: Brief Activities — The activities will be completed online.

SUMMARY:
This is a study investigating how brief online activities can influence mood and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65
* schizophrenia group - have a psychotic disorder diagnosis
* healthy control group - Do not have a current DSM-5 diagnosis via the SCID-5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire - PHQ-9 | Assessed at baseline (day 1) and after study completion, an average of a week
  Depression measure
Generalized Anxiety Disorder 7-item - GAD-7 | Assessed at baseline (day 1) and after study completion, an average of a week
  Anxiety measure
The Motivation and Pleasure Scale-Self-Report - MAP-SR | Assessed at baseline (day 1) and after study completion, an average of a week
  Negative symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request, we will share data.